CLINICAL TRIAL: NCT05024617
Title: Stage-Specific Recovery Changes in the International Classification of Functioning Components Following Conservative Rehabilitation of Trigger Finger
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cigdem Ayhan, Associate Professor (Lecturer), Hacettepe University
Other Study IDs: 16969557-437
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Trigger Finger
Keywords: trigger finger; ICF; rehabilitation; splinting
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- trigger finger stage 1-2-3: Volunteer patients between 35-65 years old diagnosed with Stage 1, Stage 2 and Stage 3 trigger finger based on the Froimson Classification were included in the study. Exclusion criteria include paediatric trigger finger, trigger thumb, concomitant de'Quervain tenosynovitis, carpal tunnel syndrome, or Dupuytren's contracture, neurological or rheumatological diseases, chronic pain syndromes, pregnancy and patients with treatment history of related finger/fingers
  Interventions: Other: conservative treatment

INTERVENTIONS:
Other: conservative treatment — All patients had rehabilitation for a total of three months, including activity modification, splinting and exercises.

SUMMARY:
The aim of this study was to determine the effectiveness of conservative rehabilitation on the multi-dimensional health components based on WHO ICF model in Stage 1, Stage 2 and Stage 3 trigger finger and to determine the functional recovery patterns of each dimension during a three-month rehabilitation period. Thirty-four patients were participated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Stage 1, Stage 2 and Stage 3 trigger finger based on the Froimson Classification

Exclusion Criteria:

* Paediatric trigger finger, trigger thumb, concomitant de'Quervain tenosynovitis, carpal tunnel syndrome, or Dupuytren's contracture, neurological or rheumatological diseases, chronic pain syndromes, pregnancy and patients with treatment history of related finger/fingers.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosed with Stage 1, Stage 2 and Stage 3 trigger finger based on the Froimson Classification
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | one month
Number of triggering (ten active fist test / 30 second active fist test) | one month
Grip strength (hand dynomometer and pinchmeter) | one month

CONTACTS AND LOCATIONS:
Overall Officials: Seda Namaldi, MSc, Principal Investigator — Hacettepe University, Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Namaldi S, Kuru CA, Kuru I. Prediction of disability in trigger finger: a cross-sectional and longitudinal study. J Hand Surg Eur Vol. 2023 Feb;48(2):131-136. doi: 10.1177/17531934221131883. Epub 2022 Nov 2. PMID 36324191